CLINICAL TRIAL: NCT06496477
Title: Light Therapy to Treat Depression in Pediatric Stem Cell Therapy Recipients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SJLIGHT; NCI-2025-03591 (Other: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2023-11-09; First posted 2024-07-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hematopoietic Stem Cell Transplant
Keywords: Depression; Sleep; Fatigue
MeSH Terms: conditions — Depression; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1-A bright blue-spectrum white light (BL (Active Comparator): Participants will receive therapy with bright blue-spectrum white light (BL) for up to thirty minutes each day for 28 days during their HSCT related hospital admission
  Interventions: Device: Ayo wearable
- Group 2- A dim blue-spectrum white light control (DL (Active Comparator): Participants will receive therapy with dim blue-spectrum white light control (DL) for up to thirty minutes each day for 28 days during their HSCT related hospital admission
  Interventions: Device: Ayo wearable

INTERVENTIONS:
Device: Ayo wearable — Primary study device - the Ayo wearable which are glasses that emit either bright blue-spectrum white light or dim blue-spectrum white light or Mini motion logger AAM-32 - an actigraphy device work during the first and last week of the study on the participants wrist throughout most of the day, measuring activity. This will be used as an indicator of sleep.

SUMMARY:
The participants are being asked to be in this clinical trial, a type of research study, because the participants are going to have a hematopoietic stem cell transplant (HSCT) in the near future. Participants that get HSCT's often get depression and/or suffer from depressive symptoms, tiredness, and sleep disturbances.

Primary Objective

To evaluate the efficacy of BL therapy for the treatment of depression in children and adolescents undergoing hematopoietic stem cell transplant.

Secondary Objectives

* To evaluate the temporal effect and magnitude of BL vs. DL therapy on depression in pediatric patients undergoing HSCT.
* To evaluate the efficacy of BL therapy for the treatment of fatigue in children and adolescents undergoing hematopoietic stem cell transplant.
* To evaluate the response of BL therapy versus DL on sleep quality.

Exploratory Objectives

* To compare incidence of positive delirium screenings between those receiving BL therapy versus DL
* To evaluate participant and caregiver perceptions of the acceptability, ease of use, and risks/benefits of the use of Light Therapy Glasses during HSCT utilizing qualitative interviews.

DETAILED DESCRIPTION:
If you decide to be in this study, you will be asked to:

* Complete some surveys before the study begins
* Take more surveys for about 4 weeks
* Wear light therapy glasses for about 30 minutes each day for about 4 weeks
* Wear a wrist monitor every day and night for the 1st and last week of the study to record your motion and sleeping habits.
* Keep a ''sleep diary" where you will mark the times that you sleep while wearing the wrist monitor.
* Complete an optional interview at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥8 to <18 years of age at the time of enrollment
* Allogeneic HSCT planned to occur between 7 and 10 days in the future from recruitment
* Patient and/or primary caregiver reads and writes in English or Spanish
* Participant/guardian is willing to sign informed consent
* Optional interview participants must be English speaking
* Baseline self-report of depressive symptoms on the PROMIS® Pediatric Depressive Symptoms v3.0 (PROMIS-PedDepSx) ≥ 55

Exclusion Criteria:

* Taking photosensitizing medications
* Total blindness / complete lack of light perception bilaterally
* Significant physiological or psychological impairment that interferes with participation
* Any patient that, in the opinion of the primary investigator is not appropriate for the study
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.
* Non-English-speaking participants will not be eligible for the optional qualitative interview
* Baseline self-report of depressive symptoms on the PROMIS® Pediatric Depressive Symptoms v3.0 (PROMIS-PedDepSx) < 55

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Depression Efficacy | Baseline
  Depressive symptoms will be assessed using the PROMIS Ped CAT v2.0 - Depressive Symptoms (Patient and Parent Proxy, though Patient report will be used for stratification and is the primary outcome measure and basis for stratification). Participants meet all eligibility criteria including baseline PROMIS scores of 55 or above will be stratified by these scores and receive weekly re-evaluation through the approximately 4-week study period.

SECONDARY OUTCOMES:
Magnitude and Temporality of Effect in Depression | Baseline
  Depressive symptoms will be assessed using the PROMIS Ped CAT v2.0 - Depressive Symptoms (Patient and Parent Proxy, though Patient report will be used for stratification and is the primary outcome measure and basis for stratification). Participants meet all eligibility criteria including baseline PROMIS scores of 55 or above will be stratified by these scores and receive weekly re-evaluation through the approximately 4-week study period. Sequential assessments are to determine the magnitude of response and time to effect of the intervention between the treatment and control conditions.
Fatigue Efficacy" (though we will also have data for magnitude and temporality given data collection is identical to the primary objective) | Baseline
  PROMIS Ped CAT v2.0 - Fatigue (Patient and Parent Proxy)
Impact on Sleep Quality" | Actigraphy devices will be worn for at least 3 days from day 0 - day 7 ± 3 days post-transplant and at least 3 days from day 21 - 28 ± 3 days post-transplant
  Participants will wear actigraphy devices (the Mini Motion Logger AAM-32) for at least 3 days from day 0 - day 7 ± 3 days post-transplant (baseline sleep measures) and at least 3 days from day 21 - 28 ± 3 days post-transplant. Actigraphy devices will be distributed at day 0 and 21 ± 3 days post-transplant and collected on day 7 and 28 ± 3 days post-transplant by a research team member while completing regularly planned study visits. During the days the device is worn, participants will do so for as much time during each day as possible, with near continuous wear being recommended. The device will collect data regarding the participants sleep minutes, sleep efficiency, defined as the percentage of time in bed spent sleeping, and wake after sleep onset, defined as minutes of awakening during a sleep phase. Data will be compared between participants receiving BL versus DL interventions in our study cohort.

OTHER OUTCOMES:
Impact on Delirium Incidence | observed for the entire duration of the intervention
  Comparison of intervention and control group rates of positive (versus negative) screening scores on the Cornell Assessment of Pediatric Delirium. This is an observational scale completed by the patient's assigned nurse near the end of each nursing shift. While the scale has a cut-off point, and the primary exploratory objective is decreased rate of positive screens (CAPD score ≥9), we will also assess the between group scores as a numeric value with a range of 0 - 32. These assessments will be used to determine any impact of the intervention to reduce positive screening rates or overall scores on the CAPD.
Participant Perceptions of Light Therapy | day 28 ± 3 days post-transplant
  An investigator created survey focused on participant and caregiver perceptions of the acceptability, ease of use, and risks/benefits will be given to all participants and/or their caregivers on day 28 ± 3 days post-transplant, and also offered to participants withdrawing from the study who have completed at least 3 light therapy sessions. Additionally, participants and/or their primary caregiver during transplant will be asked to participate in an optional qualitative interview until up to 20 interviews are completed. This interview will be focused on the same topics (perceptions of the acceptability, ease of use, and risks/benefits). This data will be analyzed using both quantitative (survey) and qualitative (interview) methods to provide deeper participant/caregiver insights into these topic areas.
Adherence | Day 1 to Day 28 ± 3 days post-transplant, once daily, between the hours of 6 AM and 3 PM CST for a period not to exceed 30 minutes.
  The light therapy devices worn from Day 1 to Day 28 ± 3 days post-transplant will automatically collect data on their use, including session initiation and length of use identified by participants opening the device's arms and initiating the session by using the connected electronic application (initiation). End-time of each session is determined by the participant closing the arms of the device, ending the session by the connected electronic application, or reaching the full 30-minute allowable length of each individual session. This maximum duration is enforced by the device manufacturer through programing prior to the devices initial use by each participant.
Adverse Effects | day 7-, 14-, 21-, and 28-days post-HSCT ± 3 days
  : Data on adverse events, both anticipated and unanticipated, will be screened for at each assessment period. Adverse events which are anticipated to occur and be potentially related to the light therapy exposure include: Headaches, Insomnia, Dry eyes, eye pain, or sensitivity to light, Fatigue, Hypomania, and Irritability.
Potential Confounding Effects | Data will be collected from chart review covering the entire duration of the intervention
  Data on number of visits with mental health providers (psychiatry and, if seen more than once for the universal pre-HSCT assessment, psychology) and exposure to medications with potential effects on mental health, as well as their intended indication will be collected from the patient's medical record. This data will be collected from the time of study enrollment until the last day of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Elliott, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols